CLINICAL TRIAL: NCT06578468
Title: Preoxygenation Using End-Tidal Oxygen for Rapid Sequence Intubation in the Emergency Department (The PREOXED Trial) - a Multicentre Stepped Wedge Cluster Randomised Control Trial
Brief Title: End-Tidal Oxygen for Intubation in the Emergency Department
Acronym: PREOXED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sydney Local Health District (Other Government)
Responsible Party: Principal Investigator, Matthew Oliver, Staff Specialist, Sydney Local Health District
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-008
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Critical Illness; Hypoxia; Respiratory Failure
Keywords: Emergency Intubation
MeSH Terms: conditions — Critical Illness; Hypoxia; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control period (No Intervention): The control period includes a period whereby clinicians will not have access to ETO2 monitoring and routine RSI practices will be documented including all study variables. At all institutions, RSI is performed in a similar manner, utilising an airway checklist. There is no 'standard operating procedure' for RSI in any of the EDs and methods, therefore, vary depending on clinician preference and the condition of the patient, however, each site is a tertiary-level, university teaching hospital and therefore clinical practice is up to date and evidence-based. Standard preoxygenation methods in the Emergency department often consist of a bag-valve mask, with or without a PEEP valve, set at 15L/min, or the use of non-invasive ventilation or a non-rebreather mask, with or without a nasal cannula, set at 15 L/min or flush rate oxygen (>40 L/min). US sites have access to high-flow (>30L/min) oxygen. This is the only difference in the preoxygenation method.
- Study period (Experimental): For all patients involved in the study, the only intervention will be the use of ETO2 to guide preoxygenation. All aspects of RSI will be at the discretion of the treating clinician including sedative/paralytic medications, positioning of the patient, preoxygenation method, intubation techniques and post-intubation sedation.
  Clinicians will be encouraged to aim for the highest ETO2 result possible with a goal of >85%. Clinicians will be able to view the ETO2 values and can decide on any changes to the preoxygenation techniques if deemed necessary. These techniques may include improved patient positioning, improved face mask seal, increased oxygen flow, length of preoxygenation time, or altering the preoxygenation device.
  Interventions: Device: End-tidal oxygen monitor

INTERVENTIONS:
Device: End-tidal oxygen monitor — The only additional equipment required for this study is the Philips™ IntelliVue G7m Gas Analyser Module 866173. This provides a non-dispersive infrared measurement of respiratory gases and a paramagnetic measurement of oxygen. At Lincoln Medical Center, the gas analyser used will be a Philips G5 gas analyser connected to a Philips Intellivue MP 70. At the University of New Mexico Medical Center, the Masimo root monitor is used.
  The gas analysers produce display waves for O2 and CO2, together with numerics for end-tidal values for O2 and CO2 and to our knowledge, there are no differences in values between the various devices used. The gas sampling occurs through a side-stream sampling tube at a rate of 200ml/min ±20 ml/min, which is either obtained from a nasal cannula in the spontaneously breathing patient or a sidestream line if connected to a BVM.
  Arms: Study period

SUMMARY:
Rapid Sequence Intubation (RSI) is a high-risk procedure in the emergency department (ED). Patients are routinely preoxygenated (given supplemental oxygen) prior to RSI to prevent hypoxia during intubation. For many years anaesthetists have used end-tidal oxygen (ETO2) levels to guide the effectiveness of preoxygenation prior to intubation. The ETO2 gives an objective measurement of preoxygenation efficacy. This is currently not available in most EDs.

This trial evaluates the use of ETO2 on the rate of hypoxia during intubation for patients in the ED.

DETAILED DESCRIPTION:
BACKGROUND AND INTRODUCTION

Rapid Sequence Intubation (RSI) is a common procedure in Emergency Departments (ED). However, it is a high-risk procedure and is associated with significant complications including hypoxia, failed intubation, hypotension, trauma and aspiration. (1-3) Specifically, hypoxia during intubation can lead to poor outcomes such as dysrhythmias, haemodynamic compromise, hypoxic brain injury and death and therefore oxygen desaturation is of primary concern during any intubation procedure. (4, 5) In order to prevent desaturation events during intubation, a number of steps are taken by clinicians. These include optimal patient positioning, adequate preoxygenation, assessment of airway anatomy and development of a detailed airway plan as well as the use of apnoeic oxygenation.(6)

Effective preoxygenation is vital to ensure that the patient does not develop hypoxia during the period between induction (administration of sedative and paralytic agents) and restoration of ventilation by successful endotracheal intubation or rescue breathing. Various methods of preoxygenation have been developed to wash the nitrogen out of the lungs (denitrogenation) which allows the functional residual capacity (FRC) to act as an oxygen reservoir during intubation, which prolongs safe apnoea time, therefore, preventing desaturation whilst an endotracheal tube (ETT) is placed.

Adequate preoxygenation is especially important for those patients at highest risk of hypoxia during the RSI. This patient group includes those with underlying lung pathology e.g. pneumonia, patients with increased metabolic demand e.g. sepsis, patients with an oxygen requirement prior to RSI, or patients with underlying conditions that predisposes to hypoxia e.g. obesity.

For many years anaesthetists have used end-tidal oxygen (ETO2) levels to guide the effectiveness of preoxygenation. ETO2 measures the exhaled oxygen concentration and is a marker of the oxygen concentration in the alveoli. Prior to induction, anaesthetists most commonly preoxygenate with a face-mask seal via either a circle circuit, Mapleson circuit, or bag valve mask. ETO2 provides an objective measurement of preoxygenation efficacy. The Difficult Airway Society guidelines suggest aiming for an ETO2 of ≥87% prior to commencing RSI.(7) ETO2 levels are not routinely measured in Emergency Departments.

Currently, it is not possible to measure the effectiveness of preoxygenation in the ED. Pulse-wave oximetry reflects peripheral oxygen saturation and not the pulmonary oxygen concentration. Therefore, to attempt to optimize preoxygenation the emergency clinician currently can only use time as a surrogate. The typically recommended duration of preoxygenation is > 3 minutes.

Recently, the investigators conducted two multi-site studies (Ethics identifier: 2019/ETH06644) that investigated the use of ETO2 in the ED.(8, 9) The first study was conducted with clinicians blinded to the ETO2 result (8). The investigators demonstrated that preoxygenation was uniformly poor with only 26% of patients achieving the required target ETO2 of ≥85%. The investigators then completed a second study where clinicians had access to ETO2 values and found that the proportion of patients reaching levels ≥85% was improved to 67% of patients. (9) The prevalence of hypoxemia (SpO2 <90%) in the group blinded to ETO2 was 18% (n=18, 95% CI: 11% to 27%) and was 8% in the group where ETO2 was available (n = 8, 95% CI: 4% to 15%). These studies indicate that the use of ETO2 may substantially improve preoxygenation in the ED and therefore reduce the risk of hypoxia.

These studies, however, were focused on preoxygenation practices and not patient-oriented outcomes (hypoxia) and were limited in design and resources. Consequently, it is still unclear whether the use of ETO2 in the ED leads to improved clinical outcomes.

RATIONALE FOR PERFORMING THE STUDY

The aim of this study is to determine the effectiveness of ETO2 monitoring in preventing desaturation for patients with a high risk of hypoxia undergoing RSI in ED.

HYPOTHESIS

The investigators hypothesise that the use of ETO2 monitoring leads to reduced rates of oxygen desaturation during the peri-intubation period compared to when it is not used.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is located in the ED resuscitation bay of the participating centre.
2. The planned procedure is orotracheal intubation using a laryngoscope and RSI technique with preoxygenation for patients who are spontaneously breathing.
3. The patient is deemed to be at a high risk of hypoxia during RSI as per the treating ED clinician, as defined by:

   * Any patient requiring any form of oxygen therapy before preoxygenation.
   * Any patient with respiratory pathology based on clinical or radiological findings. Including, but not limited to:

     * Pneumonia, pulmonary oedema, acute respiratory distress syndrome (ARDS), aspiration, pulmonary contusion from trauma, infective exacerbations of known lung disease (e.g. asthma, pulmonary fibrosis, emphysema) or pulmonary embolism (PE)
   * Any patient with high oxygen consumption. Including, but not limited to:

     * Sepsis, Diabetic ketoacidosis, alcohol or drug withdrawal, seizures, thyrotoxicosis
   * Any underlying patient condition that may predispose to hypoxemia. Including, but not limited to:

     * Obesity, pregnancy, underlying lung disease (e.g. asthma, pulmonary fibrosis, emphysema), severe injury- hypovolaemia/haemorrhage.
   * or any other patient that the treating clinician has a high concern for hypoxemia during RSI.

Exclusion Criteria:

1. Patient is known to be less than 18 years old.
2. The patient has a supraglottic device in-situ e.g iGel or LMA.
3. The patient is known to be pregnant.
4. The patient is known to be a prisoner.
5. The patient was intubated in the prehospital environment.
6. Immediate need for tracheal intubation precludes preoxygenation i.e. the patient is in cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | The time when laryngoscope first enters the mouth to 2 minutes after the endotracheal tube [ETT] is confirmed on waveform capnography
  The proportion of patients that experience oxygenation desaturation (SpO2 <93%, or >10% from baseline if SpO2 <93% at the end of preoxygenation) during the peri-intubation period

SECONDARY OUTCOMES:
Lowest oxygen saturations | The time when laryngoscope first enters the mouth to 2 minutes after the endotracheal tube [ETT] is confirmed on waveform capnography
  The lowest oxygen saturation (SpO2) during the peri-intubation period

OTHER OUTCOMES:
Time from preoxygenation to endotracheal intubation | Preoxygenation start time to endotracheal intubation confirmation
  Time from preoxygenation to endotracheal intubation
Incidence of severe oxygen desaturation (SpO2 <80%) | Induction of sedative medications and 2 minutes post ETT confirmation
  Incidence of severe oxygen desaturation (SpO2 <80%)
Incidence of very severe oxygen desaturation (SpO2 <70%) | Induction of sedative medications and 2 minutes post ETT confirmation
  Incidence of very severe oxygen desaturation (SpO2 <70%)
Incidence of the number of patients with pre-oxygenation method changes to achieve higher ETO2 in intervention arm | During preoxygenation
  Incidence in pre-oxygenation changes in method to deliver higher ETO2:
  * BVM
  * BVM+PEEP
  * HFNP
  * NIV
Incidence of the number of patients with pre-oxygenation technique changes to achieve higher ETO2 in intervention arm | During preoxygenation
  Incidence in pre-oxygenation changes in technique to deliver higher ETO2:
  * Improved mask seal
  * Increased O2 flow rate
  * Increased Preoxygenation time
Number of re-oxygenation events | During preoxygenation
  A re-oxygenation attempt is a failed first attempt at ETT placement followed by administration of an oxygen delivery device (BVM, NIV, supraglottic device) to maintain SpO2 levels
Cardiovascular complications during RSI | Induction of sedative medications and 2 minutes post ETT confirmation
  * Bradycardia (HR< 40 bpm)
  * Tachycardia (HR> 120 bpm)
  * Hypotension (SBP< 90 mm Hg or a 30mmHg reduction from baseline)
Other complications during RSI | Induction of sedative medications and 2 minutes post ETT confirmation
  Operator reported aspiration between induction and intubation Oesophageal intubation recognised after the laryngoscope blade has been removed, detected by waveform ETCO2 Cardiac arrest occurred during RSI

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Oliver, MBBS, Study Chair — Sydney Local Health District; Nick Caputo, Md, Study Chair — Lincoln Medical Center
Locations (9):
- United States (3):
  - Hennepin Medical Center, Minneapolis, Minnesota
  - University of New Mexico Medical Center, Albuquerque, New Mexico
  - Lincoln Medical Center, The Bronx, New York
- Australia (6):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Northern Beaches Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: No end date
Access Criteria: a signed data access agreement research testing a hypothesis a protocol that has been approved by an institutional review board a proposal that has received approval from the principal investigator

REFERENCES:
- [Background] Martin LD, Mhyre JM, Shanks AM, Tremper KK, Kheterpal S. 3,423 emergency tracheal intubations at a university hospital: airway outcomes and complications. Anesthesiology. 2011 Jan;114(1):42-8. doi: 10.1097/ALN.0b013e318201c415. PMID 21150574
- [Background] Bair AE, Filbin MR, Kulkarni RG, Walls RM. The failed intubation attempt in the emergency department: analysis of prevalence, rescue techniques, and personnel. J Emerg Med. 2002 Aug;23(2):131-40. doi: 10.1016/s0736-4679(02)00501-2. PMID 12359280
- [Background] Alkhouri H, Vassiliadis J, Murray M, Mackenzie J, Tzannes A, McCarthy S, Fogg T. Emergency airway management in Australian and New Zealand emergency departments: A multicentre descriptive study of 3710 emergency intubations. Emerg Med Australas. 2017 Oct;29(5):499-508. doi: 10.1111/1742-6723.12815. Epub 2017 Jun 5. PMID 28582801
- [Background] Mort TC. The incidence and risk factors for cardiac arrest during emergency tracheal intubation: a justification for incorporating the ASA Guidelines in the remote location. J Clin Anesth. 2004 Nov;16(7):508-16. doi: 10.1016/j.jclinane.2004.01.007. PMID 15590254
- [Background] Davis DP, Dunford JV, Poste JC, Ochs M, Holbrook T, Fortlage D, Size MJ, Kennedy F, Hoyt DB. The impact of hypoxia and hyperventilation on outcome after paramedic rapid sequence intubation of severely head-injured patients. J Trauma. 2004 Jul;57(1):1-8; discussion 8-10. doi: 10.1097/01.ta.0000135503.71684.c8. PMID 15284540
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Caputo ND, Oliver M, West JR, Hackett R, Sakles JC. Use of End Tidal Oxygen Monitoring to Assess Preoxygenation During Rapid Sequence Intubation in the Emergency Department. Ann Emerg Med. 2019 Sep;74(3):410-415. doi: 10.1016/j.annemergmed.2019.01.038. Epub 2019 Mar 14. PMID 30879700
- [Background] Oliver M, Caputo ND, West JR, Hackett R, Sakles JC. Emergency physician use of end-tidal oxygen monitoring for rapidsequence intubation. J Am Coll Emerg Physicians Open. 2020 Sep 28;1(5):706-713. doi: 10.1002/emp2.12260. eCollection 2020 Oct. PMID 33145509
- [Background] American College of Emergency Physicians (ACEP) Policy statement: Rapid-Sequence Intubation February 2018 [Available from: https://www.acep.org/patient-care/policy-statements/rapid-sequence-intubation/.
- [Background] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096